CLINICAL TRIAL: NCT04662515
Title: Novel Oral Anticoagulants in Oral and Maxillofacial Surgery: Impact on Bleeding Tendency, Surgical Difficulty and Post-operative Complications
Brief Title: NOACs in Oral and Maxillofacial Surgery: Impact on Post-operative Complications
Status: Completed | Type: Observational
Sponsor: Malmö University (Other)
Collaborators: Odontologisk Forskning i Region Skåne (OFRS) (Unknown)
Responsible Party: Principal Investigator, Krister Johansson, Dr Krister Johansson. Department of Oral and Maxillofacial Surgery and Oral Medicine, Faculty of Odontology, Malmö University, Malmö University
Other Study IDs: AK-BLD
Record Dates: First submitted 2020-12-04; First posted 2020-12-10 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Surgery, Oral; Hemorrhage; Postoperative Complications; Oral Surgical Procedures; Anticoagulants Causing Adverse Effects in Therapeutic Use; Anticoagulant-induced Bleeding
MeSH Terms: conditions — Hemorrhage; Postoperative Complications | interventions — Dabigatran; Rivaroxaban; apixaban; edoxaban; Warfarin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- DOAC: Information about which type of DOAC and the dose that is prescribed to the patient will be collected.
  Interventions: Procedure: Type of surgery; Drug: Dabigatran; Drug: Rivaroxaban; Drug: Apixaban; Drug: Edoxaban
- Warfarin: A PK-INR ≤3.0 retained whitin the last 24 hours have to be present for inclusion.
  Interventions: Procedure: Type of surgery; Drug: Warfarin

INTERVENTIONS:
Procedure: Type of surgery — surgical or non-surgical extraction one or more teeth
Drug: Dabigatran
  Groups: DOAC
Drug: Rivaroxaban
  Groups: DOAC
Drug: Apixaban
  Groups: DOAC
Drug: Edoxaban
  Groups: DOAC
Drug: Warfarin
  Groups: Warfarin

SUMMARY:
Aims: To investigate the incidence of bleeding complications during oral surgical procedures in patients medicated with DOACs.

To investigate the perioperative and postoperative bleeding volume during oral surgical procedures in patients medicated with DOACs.

To examine whether increased perioperative bleeding volume complicates the planned intervention, thereby prolonging the operation time.

Previous studies have shown that the incidence of healthcare-consuming bleeding complications following oral surgical procedures in patients who are prescribed warfarin is approximately 4% (9). To investigate whether the incidence is higher or lower by the intake of DOAC it is considered to be sufficient with 100 patients in each group. The groups consist of patients who are prescribed warfarin, DOACs, as well as a control group.

Hypothetical outcomes: The incidence of bleeding complications and the perioperative and postoperative bleeding volume during oral surgical procedures in patients medicated with DOACs are higher compared to patients medicated with warfarin and patients taking no anticoagulants. Increased perioperative bleeding volume complicates the planned intervention, thereby prolonging the operation time.

Clinical relevance: The study will serve as a basis for the development of treatment guidelines for patients who medicate with DOACs. If it turns out that the oral surgery procedure presents no increased risk of complications and that the bleeding volume does not complicate the surgery significantly, it may be recommended that patients who medicate with DOACs whom are in need of oral surgical procedures seek ordinary dental care.

DETAILED DESCRIPTION:
The continuous variables (amount of bleeding during surgery) will be analyzed with linear regression if they show normal distribution patterns.

The ordinal variables (postoperative bleeding complications) will be analyzed with ordinal logistic regression.

Dichotomous variables (presence of other postoperative complications) will be analyzed with logistic regression.

ELIGIBILITY:
Inclusion Criteria:

Need of dental extraction / oral surgery, and medication with:

1. warfarin or
2. DOACs or
3. no treatment or AK-platelet therapy and age-matched to group a) and b).

Exclusion Criteria:

Medication with the combination of anticoagulants and antiplatelet Ongoing drug abuse

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients referred to either the oral surgery department at Skåne University hospital or the department for Oral surgery and oral medicine, Malmö University.
  The plan is to ask all patients consecutively referred to the clinics for participation.
Sampling Method: Non-Probability Sample
Enrollment: 216 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
bleeding complication | 4 weeks postoperatively
  proportion of patients who are in need of non planned/emergency medical or dental care after tooth extraction / oral surgery because of bleeding

SECONDARY OUTCOMES:
bleeding volume | the actual time of surgery
  the amount of blood that the patient is bleeding during tooth extraction / oral surgery
surgical difficulty | the actual time of surgery
  estimation on a scale of 1-10 by the surgeon
surgery time in minutes | the actual time of surgery
proportion of other postoperative complications | 4 weeks postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Jonas P becktor, DDS, PhD, Study Director — Faculty of Odontology, Malmö University
Locations (2):
- Sweden (2):
  - Skåne University Hospital, Helsingborg
  - Department of Oral and Maxillofacial Surgery and Oral Medicine, Faculty of Odontology, Malmö University, Malmo

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Johansson K, Becktor JP, Naimi-Akbar A, Svensson PJ, Gotrick B. Continuous use of direct oral anticoagulants during and after simple and surgical tooth extractions: a prospective clinical cohort study. BMC Oral Health. 2025 Apr 12;25(1):554. doi: 10.1186/s12903-025-05949-9. PMID 40221663